CLINICAL TRIAL: NCT03153111
Title: A Multi-center, Double-blind, Placebo-controlled Phase 2b Study to Evaluate the Efficacy and Safety of Macitentan in Subjects With Heart Failure With Preserved Ejection Fraction and Pulmonary Vascular Disease
Brief Title: A Study to Evaluate Whether Macitentan is an Effective and Safe Treatment for Patients With Heart Failure With Preserved Ejection Fraction and Pulmonary Vascular Disease
Acronym: SERENADE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-055G202; 2016-003653-15 (EudraCT Number)
Record Dates: First submitted 2017-03-30; First posted 2017-05-15 (Actual); Results first posted 2022-04-04 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — macitentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Macitentan (Active Comparator): Subjects randomized to the macitentan arm receives one tablet of macitentan 10 mg every day for at least 24 to maximum 52 weeks.
  Interventions: Drug: Macitentan
- Placebo (Placebo Comparator): Subjects randomized to the placebo arm received one tablet of placebo every day for at least 24 to maximum 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Macitentan — macitentan 10 mg; film-coated tablet; oral use
  Other Names: ACT-064992
  Arms: Macitentan
Drug: Placebo — film-coated tablet (identical to the macitentan tablet); oral use
  Arms: Placebo

SUMMARY:
This is a study to evaluate whether macitentan is an effective and safe treatment for patients with heart failure with preserved ejection fraction (HFpEF) and pulmonary vascular disease.

The primary objective is to evaluate whether macitentan 10 mg reduces N-terminal pro-brain natriuretic peptide (NT-pro-BNP) as compared to placebo in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Signs or symptoms of Heart Failure (HF) (NYHA FC I I and II I ) requiring treatment with at least one oral diuretic (any type)
* Left ventricular ejection fraction (LVEF) ≥ 40% (by echocardiography at Screening)
* Structural heart disease consistent with heart failure with preserved ejection fraction (HFpEF) established by echocardiography at Screening
* Elevated NT-proBNP
* Pulmonary vascular disease or right ventricular dysfunction

Exclusion Criteria:

* Any prior valid measurement of LVEF < 40%. An echocardiogram is considered valid if its quality is sufficient to allow accurate assessment of LVEF and if it is reflective of the true status of the subject
* Cardiovascular co-morbidities (e.g., significant unrepaired structural valvular heart disease; acute coronary syndrome, coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI) within 3 months of Screening; uncontrolled heart rate from atrial fibrillation or atrial flutter, history of serious life-threatening or hemodynamically significant arrhythmia; history of or anticipated heart transplant or ventricular assist device implantation, etc)
* Systolic blood pressure (SBP) ≥ 180 mmHg, or diastolic blood pressure (DBP) ≥ 110 mmHg during Screening
* Hemoglobin < 100g/L (< 10 g/dl) at Screening
* Significant parenchymal lung disease (e.g., severe COPD, moderate or severe restrictive lung disease, diffuse interstitial fibrosis or alveolitis, pulmonary thromboembolism)
* Severe renal dysfunction with an estimated Glomerular Filtration Rate (eGFR) < 30 mL/min per 1.73 m2
* Severe hepatic impairment, e.g., Child Pugh Class C

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (95):
- United States (24):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Cedars Sinai Heart Institute, Beverly Hills, California
  - Sharp Memorial Hospital, San Diego, California
  - Harbor Ucla Medical Center, Torrance, California
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University Of Iowa - Hospitals & Clinics, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School Of Medicine, St Louis, Missouri
  - Weill Cornell Medicine, New York, New York
  - Peak Clinical Trials, Apex, North Carolina
  - University of North Carolina (UNC) - School of Medicine, Chapel Hill, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Allegheny, Pittsburgh, Pennsylvania
  - Vascular Medicine Institute University Of Pittsburgh, Pittsburgh, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - North Dallas Research Associates, McKinney, Texas
  - Baylor Scott and White Research Institute, Temple, Texas
  - Inova Heart and Vascular Institute, Falls Church, Virginia
  - MultiCare Health System, Tacoma, Washington
  - Aurora Saint Lukes Medical Center, Milwaukee, Wisconsin
- Argentina (4):
  - Centro Médico Dra. De Salvo, Buenos Aires
  - CCBR - Buenos Aires - AR, Buenos Aires
  - Clinica Adventista Belgrano, CABA
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata
- Medizinische Universitaet Wien, Vienna, Austria
- Brazil (5):
  - Maestri E Kormann Consultoria Médico- Científica Ltda, Blumenau
  - Rede D or Sao Luiz S A Hospital do Coracao do Brasil, Brasília
  - Instituto de Pesquisa Clinica de Campinas, Campinas
  - Instituto do Coracao de Marília, Marília
  - Instituto de Moléstias Cardiovasculares Tatuí, Tatuí
- Bulgaria (4):
  - Specialized Hospital for Active Treatment in Cardiology - Pleven, Pleven
  - Diagnostic Consulting Center I Sliven, Sliven
  - Multiprofile Hospital for Active Treatment - National Heart Hospital, Sofia
  - University Multiprofile Hospital for Active Treatment- UMHAT Sveta Anna AD, Sofia
- Czechia (5):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - University Hospital Plzeň-Lochotín, Pilsen
  - General University Hospital II.department of Internal Medicine-cardiology and angiology, Prague
  - IKEM, Prague
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus
  - Bispebjerg Og Frederiksberg Hospital, Copenhagen
  - Sydvestjysk Sygehus, Esbjerg
- France (5):
  - Hopital Henri Mondor, Créteil
  - CHU de Grenoble Hopital Albert Michallon, Grenoble
  - Hopital de Bicetre, Le Kremlin-Bicêtre
  - Hopital Cardiologique, Lille
  - CHU Rouen Hopital Charles Nicolle, Rouen
- Germany (7):
  - Charite Universitatsmedizin Berlin Campus Virchow Klinikum, Berlin
  - Universitatsklinikum Bonn, Bonn
  - Herzzentrum Uniklinik Köln Klinik III für Innere Medizin, Cologne
  - Universitätsklinikum Carl Gustav Carus Medizinische Klinik und Poliklinik 1-Pneumologie, Dresden
  - Universitaetsklinikum Giessen, Giessen
  - Universitaetsklinikum Schleswig Holstein Campus Kiel, Kiel
  - Klinikum Würzburg Mitte gGmbH Standort Missioklinik, Würzburg
- Hungary (3):
  - Budai Irgalmasrendi Korhaz, Budapest
  - Semmelweis Egyetem Varosmajor Sziv es Ergyogyaszati Klinika, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
- Israel (8):
  - Barzilai Medical Center, Ashkelon
  - Hillel Yaffe Medical Center, Hadera
  - Bnai Zion Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center Beilinson Campus, Petah Tikva
  - Kaplan Medical Center, Rehovot
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Krakowski Szpital Specjalityczny im Jana Pawla II Oddzial Kliniczny Chorob Serca i Naczyn, Krakow
  - Wojewodzki Szpital Specjalistyczny im Stefana Kardynala Wyszynskiego SPZOZ, Lublin
  - 4 Wojskowy Szpital Kliniczny Z Poliklinika SP ZOZ, Wroclaw
- Romania (4):
  - Institutul de urgenta pentru Boli Cardiovasculare Prof. Dr. C.C. Iliescu, Bucharest
  - Cardiomed, Craiova
  - SAL MED Pitesti, Piteşti
  - Cmi Dr Podoleanu Cristian, Târgu Mureş
- Russia (8):
  - Federal State Budget Scientific Institution, Kemerovo
  - Krasnodar Regional Clinical Hospital, Krasnodar
  - Moscow City Clinical Hospital No.51, Moscow
  - National Medical Research Center of Cardiology of MoH of Russian Federation, Moscow
  - Federal State Budgetary Institution, Saint Petersburg
  - State Healthcare Institution, Regional Clinical Cardiology Dispensary, Saratov
  - State Autonomous Healthcare Institution Of Yaroslavl Region, Yaroslavl
  - Ekaterinburg City Clinical Hospital #14, Yekaterinburg
- Spain (5):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario La Fe, Valencia
- Sahlgrenska Universitetsjukhuset, Gothenburg, Sweden
- United Kingdom (4):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Castle Hill Hospital, Cottingham
  - Royal Free Hospital, London
  - Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah SJ, Bonderman D, Borlaug BA, Cleland JGF, Lack G, Lu W, Voors AA, Zannad F, Gladwin MT. Macitentan for Heart Failure With Preserved or Mildly Reduced Ejection Fraction and Pulmonary Vascular Disease: Results of the SERENADE Randomized Clinical Trial and Open-Label Extension Study. Circ Heart Fail. 2025 Mar;18(3):e011381. doi: 10.1161/CIRCHEARTFAILURE.123.011381. Epub 2025 Mar 11. PMID 40066571

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 143 enrolled participants, 1 participant was randomized by mistake and did not receive any dose of study drug. 142 participants received the study drug and were analyzed.
Groups:
- Macitentan: Participants received macitentan 10 milligrams (mg) tablet orally once a day starting from Day 1 up to Week 52.
- Placebo: Participants received placebo tablet orally once a day starting from Day 1 up to Week 52.
Period: Overall Study
Arm/Group | Macitentan | Placebo
Started | 71 | 71
Completed | 60 | 62
Not Completed | 11 | 9
Not completed — Death | 2 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 5 | 1
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis population includes full analysis set (FAS) which included participants randomized to double-blind study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Macitentan | Placebo | Total
Number analyzed (Participants) | 71 | 71 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.9 (10.11) | 74.2 (8.25) | 73.6 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 41 | 87
  Male | 25 | 30 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 69 | 67 | 136
  Unknown or Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Black or African American | 3 | 1 | 4
  White | 68 | 67 | 135
  Other | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 0 | 1 | 1
  AUSTRIA | 1 | 1 | 2
  BRAZIL | 2 | 0 | 2
  BULGARIA | 4 | 6 | 10
  CZECH REPUBLIC | 2 | 1 | 3
  DENMARK | 0 | 2 | 2
  FRANCE | 2 | 4 | 6
  GERMANY | 9 | 4 | 13
  HUNGARY | 3 | 6 | 9
  ISRAEL | 13 | 14 | 27
  POLAND | 3 | 5 | 8
  ROMANIA | 5 | 2 | 7
  RUSSIAN FEDERATION | 9 | 11 | 20
  SPAIN | 0 | 1 | 1
  SWEDEN | 1 | 1 | 2
  UNITED KINGDOM | 4 | 1 | 5
  UNITED STATES | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percent of Baseline N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) Assessed at Week 24
Description: Percent of baseline NT-proBNP assessed at Week 24 was reported. Percent of baseline is calculated as the ratio of the Week 24 NT-proBNP value over baseline value, expressed in percentage. NT-proBNP is one of the best established cardiovascular response markers among all available surrogates in heart failure (HF).
Time Frame: Week 24
Population: Full analysis set (FAS) included participants which were randomized to double-blind study treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of baseline NT-proBNP
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 71 | 71
percentage of baseline NT-proBNP | 108.39 (0.65) | 106.27 (0.55)
Statistical Analysis 1: Comparison: Macitentan vs Placebo; Test type: Superiority; p = 0.7923, ANCOVA; Geometric mean ratio = 1.02, 90% CI 2-sided [0.88 to 1.19]

2. Secondary Outcome: Change From Baseline to Week 24 in the Clinical Summary Score Assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) Score
Description: The KCCQ is a validated health related quality of life measure for heart failure. The KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Clinical summary score is one of the quality of life variable of interest derived from KCCQ. Clinical summary score is the mean of domains: physical limitations score (6 items) and total symptom score (2 items [symptoms frequency and symptom burden]). The score is calculated by summing domain responses and then transforming scores to a 0-100 unit scale with higher scores indicating better health status.
Time Frame: Baseline to Week 24
Population: FAS included participants which were randomized to double-blind study treatment. Here, 'N' (number of participants analyzed) specifies all participants who were evaluated for this outcome measure (OM).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 69 | 71
score on a scale | -2.37 (16.12) | 0.89 (17.72)
Statistical Analysis 1: Comparison: Macitentan vs Placebo; Test type: Superiority; p = 0.2172, ANCOVA; Least square mean difference = -3.50, 90% CI 2-sided [-8.17 to 1.17], Standard Error of Mean 2.82

3. Secondary Outcome: Change From Baseline to Week 24 in Accelerometer-assessed Proportion of Time Spent in Light to Vigourous Physical Activity
Description: Physical activity is assessed by accelerometer as the proportion of time spent in light to vigorous physical activity based on a threshold of greater than (>)100 activity counts per minute and expressed as change from baseline to Week 24.
Time Frame: Baseline to Week 24
Population: FAS included participants which were randomized to double-blind study treatment. Here, 'N' (number of participants analyzed) specifies all participants who were evaluated for this OM.
Measure: Mean (Standard Deviation); unit: proportion of time spent
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 30 | 31
proportion of time spent | -0.024 (0.084) | -0.005 (0.098)
Statistical Analysis 1: Comparison: Macitentan vs Placebo; Test type: Superiority; p = 0.3665, ANCOVA; Least square mean difference = -0.02, 90% CI 2-sided [-0.05 to 0.02], Standard Error of Mean 0.02

4. Secondary Outcome: Number of Participants With Worsening of Heart Failure (WHF) Events Over 52 Weeks
Description: Number of participants with WHF events were reported. A WHF event includes HF death, hospitalization for WHF or an urgent visit for WHF.
Time Frame: Weeks 16, 24, 36, 52
Population: FAS included participants which were randomized to double-blind study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 71 | 71
Participants
  Week 16 | 12 | 5
  Week 24 | 14 | 6
  Week 36 | 17 | 9
  Week 52 | 18 | 13

ADVERSE EVENTS:
Time Frame: Up to 17 months
Description: Safety analysis set include all participants from full analysis set who received at least one dose of double-blind study treatment.
Arm/Group | Macitentan | Placebo
All-Cause Mortality (participants affected / at risk) | 2/71 | 5/71
Serious Adverse Events (participants affected / at risk) | 29/71 | 23/71
Other Adverse Events (participants affected / at risk) | 57/71 | 54/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan (N=71) | Placebo (N=71)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypoplastic Anaemia (Blood and lymphatic system disorders) | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0
Acute Left Ventricular Failure (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0
Acute Right Ventricular Failure (Cardiac disorders) | 0 | 0
Angina Pectoris (Cardiac disorders) | 1 | 1
Angina Unstable (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular Block Complete (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 1
Cardiac Failure Acute (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 5 | 0
Chronic Right Ventricular Failure (Cardiac disorders) | 1 | 0
Left Ventricular Failure (Cardiac disorders) | 3 | 2
Right Ventricular Failure (Cardiac disorders) | 6 | 6
Sinus Node Dysfunction (Cardiac disorders) | 0 | 1
Diabetic Retinopathy (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 1
Oedema Peripheral (General disorders) | 0 | 1
Congestive Hepatopathy (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 3
Pneumonia Viral (Infections and infestations) | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0
Pyelonephritis Acute (Infections and infestations) | 1 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 | 0
Sepsis (Infections and infestations) | 0 | 0
Septic Shock (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 2
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0
Ammonia Increased (Investigations) | 1 | 0
Blood Lactic Acid Increased (Investigations) | 0 | 1
Haemoglobin Decreased (Investigations) | 1 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0
Fluid Retention (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Superficial Spreading Melanoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2
Oliguria (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 1 | 0
Uterine Polyp (Reproductive system and breast disorders) | 1 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 0
Hypertension (Vascular disorders) | 0 | 0
Hypotension (Vascular disorders) | 0 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan (N=71) | Placebo (N=71)
Anaemia (Blood and lymphatic system disorders) | 5 | 3
Blood Loss Anaemia (Blood and lymphatic system disorders) | 2 | 1
Hypochromic Anaemia (Blood and lymphatic system disorders) | 2 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 4 | 1
Normocytic Anaemia (Blood and lymphatic system disorders) | 2 | 1
Angina Pectoris (Cardiac disorders) | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 4 | 5
Atrial Flutter (Cardiac disorders) | 2 | 1
Cardiac Failure Congestive (Cardiac disorders) | 3 | 1
Left Ventricular Failure (Cardiac disorders) | 5 | 0
Palpitations (Cardiac disorders) | 0 | 2
Right Ventricular Failure (Cardiac disorders) | 5 | 2
Hypothyroidism (Endocrine disorders) | 1 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 3 | 1
Fatigue (General disorders) | 5 | 6
Non-Cardiac Chest Pain (General disorders) | 1 | 2
Oedema Peripheral (General disorders) | 9 | 4
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Bronchitis (Infections and infestations) | 4 | 2
Conjunctivitis (Infections and infestations) | 2 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1
Pneumonia (Infections and infestations) | 2 | 5
Respiratory Tract Infection Viral (Infections and infestations) | 2 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 4
Urinary Tract Infection (Infections and infestations) | 2 | 5
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 4
Alanine Aminotransferase Increased (Investigations) | 2 | 1
Blood Creatinine Increased (Investigations) | 3 | 2
Blood Potassium Increased (Investigations) | 1 | 2
Blood Urea Increased (Investigations) | 4 | 1
Blood Uric Acid Increased (Investigations) | 1 | 3
Brain Natriuretic Peptide Increased (Investigations) | 0 | 2
Glomerular Filtration Rate Decreased (Investigations) | 2 | 2
Haemoglobin Decreased (Investigations) | 3 | 3
Weight Increased (Investigations) | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Fluid Retention (Metabolism and nutrition disorders) | 2 | 1
Gout (Metabolism and nutrition disorders) | 6 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Iron Deficiency (Metabolism and nutrition disorders) | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Cerebral Ischaemia (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 3 | 3
Headache (Nervous system disorders) | 4 | 1
Lethargy (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 1 | 2
Acute Kidney Injury (Renal and urinary disorders) | 5 | 2
Renal Failure (Renal and urinary disorders) | 2 | 4
Renal Impairment (Renal and urinary disorders) | 5 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Hypertension (Vascular disorders) | 2 | 2
Hypotension (Vascular disorders) | 3 | 3

LIMITATIONS AND CAVEATS:
Recruitment was stopped prematurely in December 2019 due to slow enrollment which resulted in an underpowered study and impacted the meaningful interpretation of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT03153111/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT03153111/SAP_001.pdf